CLINICAL TRIAL: NCT03349931
Title: Prospective Multicenter Evaluation of the MycoGenie Kit for the Diagnosis of Invasive Aspergillosis in Hematological Patients
Brief Title: Prospective Multicenter Evaluation of the MycoGenie Kit for the Diagnosis of Invasive Aspergillosis
Acronym: MYCOGENIE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société ADEMTECH SA (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: K-170102; 2017-A01518-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Invasive Aspergillosis in Patients With Onco-haematological Diseases
Keywords: Aspergillosis,; qPCR; allogenic haemopoietic stem-cell transplantation; leukemia
MeSH Terms: conditions — Aspergillosis; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human sera (serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematological patients: Hematological patients at high risk for invasive aspergillosis
  Interventions: Diagnostic Test: DNA extraction and detection of Aspergillus fumigatus in serum samples

INTERVENTIONS:
Diagnostic Test: DNA extraction and detection of Aspergillus fumigatus in serum samples — Performances diagnostic test of the real-time PCR ADEMTECH kit of DNA extraction and detection of Aspergillus fumigatus in serum samples in patients at high-risk for invasive aspergillosis (IA).

SUMMARY:
The purpose of this study is to evaluate the performances of the real-time PCR ADEMTECH kit of DNA extraction and detection of Aspergillus fumigatus in serum samples in patients at high-risk for invasive aspergillosis (IA). DNA detection will be associated with detection of TR34/L98H mutations in cyp51A gene, which confer azole resistance.

DETAILED DESCRIPTION:
Accurate diagnosis of invasive pulmonary aspergillosis (IPA) in patients at high risk of invasive fungal infection remains challenging due to difficulties in differentiating IPA from pulmonary infections caused by other molds or bacteria on clinical and radiological grounds. Therefore, culture-based microbiological diagnosis is of primary importance but requires semi-invasive or invasive procedures, such as bronchoalveolar Lavage (BAL) or computed-tomography (CT)-guided needle biopsy.

Alternate diagnostic methods include the detection of biomarkers, such as fungal antigens (Aspergillus galactomannan [GM]) or DNA released by Aspergillus hyphae in host tissues. These biomarkers are well recognized as early IPA predictors Recently, several clinical evaluations to detect Aspergillus DNA, either in respiratory or in blood-based samples, have clearly shown the diagnostic value of this biomarker. In addition, methodological recommendations have been established for PCR protocols, and different standardized Aspergillus quantitative PCR (qPCR) kits have been commercialized. These recent advances show that PCR is now mature for routine use in clinical settings.

Another issue is the emergence of aspergillosis due to azole-resistant isolates. Acquired azole resistance in A. fumigatus has been reported since 1997 and has emerged in many countries, particularly in Europe, as well as on other continents. In some instances, acquired resistance may be driven by antifungal selection in patients receiving long-term therapy. Nevertheless, it seems that many azole-resistant strains originated in the environment due to selection by azole fungicides used in agriculture. Azole resistance in A. fumigatus is associated mainly with mutations in the cyp51A gene, and among several mutations described, the most frequent is the mutation comprising a 34-bp tandem repeat (TR34) and the L98H alteration. Since azoles are the recommended first-line treatment for IPA, the emergence of azole resistance is worrisome and has been shown to be associated with an increased rate of clinical failure. For these reasons, routine antifungal susceptibility testing of clinical isolates has been recommended recently. Nevertheless, isolates are not always retrieved in culture, particularly for patients with hematological malignancies. Therefore, molecular detection of resistance may be a major advance for the management of patients with invasive aspergillosis.

The aim of this study will be to validate the new MycoGENIE A. fumigatus real-time PCR kit and to evaluate its performance on clinical samples for the detection of A. fumigatus and its azole resistance. This multiplex assay detects DNA from the A. fumigatus species complex by targeting the multicopy 28S rRNA gene and specific TR34 and L98H mutations in the single-copy number cyp51A gene of A. fumigatus.

The study will be performed in hematological patients with high-risk of developping IA during the course of chemotherapy. In these patients, bi-weekly detection of GM is routinely performed in all centers in France. The PCR will be performed on the samples used for GM detection. DNA will be extracted according to the manufacturer's protocol, using the MycoGENIE kit for AutoMag solution. Real-time PCR for the detection of A. fumigatus DNA will be performed using the MycoGENIE A. fumigatus real-time PCR kit (Ademtech, Pessac, France).

AI will be defined as proven or probable aspergillosis, according to EORTC criteria.

For each patient, clinical data will be collected in each center. These data include: EORTC classification, type and duration of antifungal treatments, results of GM tests, results of mycological cultures, and results of PCR tests (positivity and Ct values). For each patient a case report form (CRF) will be filled and transfered to the investigating center for analysis. Sensitivity, specificity, PPV and NPV of the PCR test will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients (≥ 18 years) hospitalized in onco hematologic unit or in hematopoietic stem cell transplantation (HSCT) unit
2. Patients with acute leukemia undergoing induction for AML, ALL, chimotherapy with neutopenia >10 days or Patients undergoing allogeneic stem cell chemotherapy transplantation
3. Patients with biweekly screening for GM detection in serum

Exclusion Criteria:

1. Patient < 18 years-old (minor)
2. Informed consent not available
3. Patient without affiliation to French social insurance
4. Patient without biweekly screening for GM detection in serum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematological patients at high risk for invasive aspergillosis, who can be classified according to EORTC criteria
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Performance of PCR for Aspergillosis diagnosis | 6 months
  Determination of the performances (Sensitivity, specificity, PPV and NPV) of the kit

SECONDARY OUTCOMES:
Detection of azole resistance | 6 months
  Detection of TR34 and L98H mutations in the A. fumigatus single-copy number gene cyp51A.

CONTACTS AND LOCATIONS:
Overall Officials: Eric DANNAOUI, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marie-Elisabeth BOUGNOUX, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (6):
- France (6):
  - Hôpital Necker - Enfants maladies (AP-HP), Paris, Paris
  - CHU Bordeaux, Groupe hospitalier, Bordeaux
  - CHU de DIJON, Hôpital du bocage, Dijon
  - CHRU de Lille, Hôpital Claude Huriez, Lille
  - CHU de Nantes, Hôpital de Moncousu, Nantes
  - CHU de RENNES, hôpital de Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suarez F, Lortholary O, Buland S, Rubio MT, Ghez D, Mahe V, Quesne G, Poiree S, Buzyn A, Varet B, Berche P, Bougnoux ME. Detection of circulating Aspergillus fumigatus DNA by real-time PCR assay of large serum volumes improves early diagnosis of invasive aspergillosis in high-risk adult patients under hematologic surveillance. J Clin Microbiol. 2008 Nov;46(11):3772-7. doi: 10.1128/JCM.01086-08. Epub 2008 Sep 24. PMID 18845828
- [Background] Dannaoui E, Gabriel F, Gaboyard M, Lagardere G, Audebert L, Quesne G, Godichaud S, Verweij PE, Accoceberry I, Bougnoux ME. Molecular Diagnosis of Invasive Aspergillosis and Detection of Azole Resistance by a Newly Commercialized PCR Kit. J Clin Microbiol. 2017 Nov;55(11):3210-3218. doi: 10.1128/JCM.01032-17. Epub 2017 Aug 16. PMID 28814586